CLINICAL TRIAL: NCT06109025
Title: Improvement of Motor Imaginative Ability Through Functional Electrical Stimulation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IO 2/2023
Record Dates: First submitted 2023-10-16; First posted 2023-10-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Electrode Site Reaction; Therapy, Directly Observed
MeSH Terms: conditions — Directly Observed Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): The sample will be composed mainly, but not exclusively, of adults of legal age, belonging to the group of university students.
  Interventions: Combination Product: FESIA GRASP; Combination Product: VIRTUAL REHAB
- CONTROL GROUP (Active Comparator): The sample will be composed mainly, but not exclusively, of adults of legal age, belonging to the group of university students.
  Interventions: Combination Product: GLOBUS ELITE

INTERVENTIONS:
Combination Product: FESIA GRASP — The Fesia Grasp device is based on the superficial electrical stimulation of the forearm musculature to provoke flexion and extension movements of the wrist, thumb, index finger and fingers 3, 4 and 5.
  Arms: EXPERIMENTAL GROUP
Combination Product: VIRTUAL REHAB — VirtualRehab is a therapeutic physical rehabilitation tool that uses virtual reality to provide therapy for patients with neurological or musculoskeletal disorders; providing a wide range of activities designed to improve mobility, coordination and strength.
  Arms: EXPERIMENTAL GROUP
Combination Product: GLOBUS ELITE — is an electro-stimulator designed for sport and fitness, but with special attention also for beauty treatments thanks to the new sequential stimulation currents, excellent for their draining effects.
  Arms: CONTROL GROUP

SUMMARY:
This is a experimental, randomised, parallel-group, clinical study.

A sample of university students will be divided into 4 groups, where one of them will act as a control group (no intervention), and the other three will undergo hand training with two different types of functional electrical stimulation devices and a final group will receive hand training with video games.

Inter-group analyses will be performed before the start of the training (pre-intervention), after the end of the programme (post-intervention), and three weeks after the end of the programme (follow-up assessment). Intra-group analyses will also be carried out to check whether the training has led to an improvement in the quality of motor imagination, as well as an improvement in manual dexterity in each of the groups.

In order to carry out the project, a collaboration agreement will be signed with the company FESIA

TECHNOLOGY S.L, which will provide a FESIA GRASP device for the study, as well as the consumables (electrodes).

DETAILED DESCRIPTION:
The study aims to answer the research question:

P: healthy adults I: FES and, FES multi-field. C: video games O: Motor imagination, strength, manual dexterity.

The aim is to compare different tools in a population sector to see if there is an improvement in motor skills through the use of these devices.

General objective: To test the effects of functional electrical stimulation and virtual reality with respect to motor imagination, strength and manual dexterity.

Secondary objectives:

To find out whether functional electrical stimulation improves motor imagination, both kinaesthetic and visual, as well as manual dexterity and strength.

To find out if an intervention based on the use of virtual reality improves motor imagination, both kinaesthetic and visual, as well as manual dexterity.

To test whether there are differences between functional electrical stimulation, multi-field functional electrical stimulation and virtual reality in terms of visual motor imagination, kinaesthetic imagination and manual dexterity.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age and sign the informed consent form.
* Not suffer from any pathology in the upper limb such as tendinitis, oedema, fractures, etc.
* Intact skin (no breaks, scratches, cuts, and other superficial or deep injuries) on the arm where the devices will be placed if applicable.

Exclusion Criteria:

* Severe medical problems.
* Use of a pacemaker.
* Pregnancy.
* Cutaneous neuropathies.
* Presence of other neuromuscular pathologies.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Nine Hole Peg Test | 1 WEEK
  The Nine Hole Peg Test (NHPT) (Mathiowetz et al, 1985), consists of a manual test, in which the subject must place 9 pegs in their corresponding 9 holes, and remove them again, the variable measured being the time it takes to carry out the whole process.
Box and Block: | 1 WEEK
  The Box and Block scale is a tool with standardised dimensions and materials. It specifies that the subject should sit in front of a rectangular box with his or her hands next to it. The box is constructed of wood with a base 53.7 cm wide and 25.4 cm long; it is divided into two square compartments of 25.4 cm each side separated by a 15.2 cm high divider; both compartments are padded in order to reduce noise during testing. The test contains 150 cube-shaped wooden blocks of 2.5 cm on each side. The number of blocks the subject has carried from one compartment to the other with each hand in one minute of time is to be recorded. Higher scores indicate better manipulative skills.
Jamar hand-held dynamometer | 1 WEEK
  The Jamar hand dynamometer is used to measure grip strength in the hand, allowing the force exerted by the individual to be converted into a numerical reading. The subject is asked to grip the device and is instructed to perform the maximum sustained contraction. The force is recorded in kilograms.
Movement imagery Questionnaire, revisado (MIQ-RS) | 1 WEEK
  The MIQ-RS questionnaire (Gregg et al, 2010) consists of 2 subscales, one visual and one kinaesthetic, of 7 items each, each item being scored on a 7-point Likert scale (the higher the score, the easier it is to imagine). For all items, the user is asked to perform a certain motor act (only once), to return to the starting position, and then to imagine it. When scoring the visual scale, the participant is asked to generate an image "as if they could see themselves" doing the gesture, while the kinaesthetic scale asks them to "recall the sensation of the movement".
  The administration manual specifies that the visual and kinaesthetic items will not be administered consecutively, but are randomly altered to avoid bias.
  The minimum values are 14, and the maximum values are 98 (minimum 7 and maximum 49 for the subscales).
Chronometry | 1 WEEK
  Chronometry is defined as the temporal congruence between an executed motor act and the same imagined act.
  In this case, the NHPT itself is proposed as the motor act executed. So, once administered to obtain the test variable (time taken to perform), the participant will be asked to imagine the performance of the test, and both measures will be timed.

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Santamaría Vázquez, PhD, Principal Investigator — University of Burgos
Locations (1):
- Olalla Saiz Vazquez, Burgos, Spain

IPD SHARING:
Plan to Share IPD: Yes
All participants will receive an informed consent form explaining the study to be carried out and the data to be used.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available throughout the intervention with participants for 3 months.
Access Criteria: Being a study participant: each participant will be provided with a password to access their informed consent and the research protocol.

REFERENCES:
- [Derived] Santamaria-Vazquez M, Ortiz-Huerta JH, Martin-Odriozola A, Saiz-Vazquez O. Improvement of Motor Imagination and Manual Ability Through Virtual Reality and Selective and Nonselective Functional Electrical Stimulation: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Nov 22;13:e63329. doi: 10.2196/63329. PMID 39576986

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT06109025/Prot_SAP_ICF_000.pdf